CLINICAL TRIAL: NCT07114887
Title: Enhancing Vocational Support With a Virtual Reality Vocational Skills Building Application: Piloting VR4VR
Brief Title: Virtual Reality for Vocational Recovery
Acronym: VR4VR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Orygen (Other)
Collaborators: TAL Community Foundation (Unknown); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ORY-P05-24-31
Record Dates: First submitted 2025-07-08; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual reality for vocational recovery (Experimental): Within standard vocational care, young people will receive a three-session (optional 4th) virtual reality training intervention to address key challenges associated with educational and employment attainment and maintenance.
  Session 1: Approaching potential employers Session 2: Asking for reasonable adjustments Session 3: Managing customers
  Interventions: Behavioral: Virtual reality for vocational recovery

INTERVENTIONS:
Behavioral: Virtual reality for vocational recovery — Intervention is an immersive virtual reality (VR) intervention, delivered through a VR headset, supported by a trained vocational specialist. Intervention content was co-designed with young people with mental health and vocational challenges, and vocational specialists with experiencing supporting this population. Content was guided by goals of vocational programs, including Individual Placement and Support.
  Other Names: VR4VR

SUMMARY:
Unemployment is higher among young people who experience mental ill-health compared to the general population. This can have a lasting impact on young people, many of whom are highly motivated to gain employment and education. There are many challenges to seeking, gaining, and maintaining employment for young people. To address these challenges and help young people meet their employment and education goals, investigators have developed a VR intervention to support vocational skill building. The aim of the current study is to evaluate the feasibility, acceptability, and safety, of the Virtual Reality for Vocational Recovery (VR4VR) intervention. A small group of vocational specialists will support up to 20 young people with their vocational outcomes using VR4VR over a 3-6week period. Both young people and specialists will complete questionnaires related to acceptability of the intervention, including qualitative interviews. Data on feasibility and safety will also be collected. Results will inform whether VR is feasible, acceptable, and safe to support vocational outcomes within vocational services that support young people with mental health difficulties, potentially supporting further intervention development and larger trials.

ELIGIBILITY:
A young person participant will be considered eligible for inclusion in this study if:

1. They are aged 18-25 seeking vocational support at participating vocational support programs
2. Have a named care-coordinator or key worker
3. Comfortable using a VR headset
4. Consent to recording of interview for transcription

Exclusion Criteria:

1. They lack fluency in English (spoken and written), since this is required to understand participate in the VR intervention;
2. They have a known diagnosis of a moderate intellectual disability, due to some of the content delivered during the intervention requiring a certain level of understanding.
3. As the therapy uses audio and visual means of communication, participants with impairments so severe that they cannot hear instructions, or are unable to see the virtual reality environments, cannot participate. Mild impairments can be accommodated, as sound volume can be turned up, and the Meta Quest headband is used to comfortably use glasses with the headset.

A vocational specialist or staff participant will be considered eligible for inclusion in this study if:

1. Presently work within a vocational program and hold a caseload of young people
2. Have worked with at least 5 young people within a vocational intervention.
3. Sufficient command of the English language
4. Consent to audio recording of interview

No exclusion criteria

A staff participant will be considered eligible for inclusion in this study if:

1. Presently work within a role supporting a vocational program
2. Sufficient command of the English language
3. Consent to audio recording of interview

No exclusion criteria

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - recruitment rates | 6 months post intervention commencement
  Rates of recruitment for the study (young people and vocational and service staff) based on an audit of study enrolment
Acceptability | 6 weeks post intervention commencement
  Acceptability as measured by the Theoretical Framework of Acceptability Measure delivered to young people and vocational specialists. Total mean score across the 7 TFA items will be reported, on a scale of 1 to 5, with 5 indicating greater acceptability.
Safety - adverse events | 6 weeks post intervention commencement
  The number of serious adverse events specifically related to the intervention or trial
Feasibility - consent rates | 6 months post intervention commencement
  Rates of consent for the study (young people and vocational and service staff) based on an audit of consent logs

SECONDARY OUTCOMES:
Feasibility - attendance rates of assessments and sessions | 6 weeks post intervention commencement
  Via audit of attendance logs
Feasibility - delivery of VR4VR | 6 months post intervention commencement
  Proportion of trained vocational specialists who use the intervention during the trial period
Feasibility - VR utilisation | 6 months post intervention commencement
  Proportion of sessions within the intervention period in which VR was used within intervention sessions.
Acceptability - cybersickness | 6 weeks post intervention commencement
  Cybersickness as measured by the Simulator Sickness Questionnaire. 16 items across three domains, nausea, Oculomotor and disorientation are summed to produce a total score. Items are scored on a scale from 0 to 3, with a higher score indicating greater cybersickness symptoms.
Acceptability - VR presence | 6 weeks post intervention commencement
  Sense of 'being there' within the VR environment measured using the Igroup Presence Questionnaire. Total score is calculated by summing all items. Items are rated on a scale of -3 to 3, with a higher scoring indicating greater sense of presence.
Effectiveness - Social and occupational functioning | 6 weeks post intervention commencement
  Young person functioning measured by the single item social and occupational functioning scale, ranging from 0 to 100, with lower scores indicating poorer functioning.
Effectiveness - Occupational self-efficacy | 6 weeks post intervention commencement
  Young person self-efficacy around employment measured by occupational self-efficacy scale. Items rated on a scale tanging from 1 to 6, with higher vales reflecting higher occupational self-efficacy.
Effectiveness - General self-efficacy | 6 weeks post intervention commencement
  Young person self-efficacy using the general self-efficacy scale, to assess an individual's perceived generalised capabilities to respond to a variety of challenges and situations. Scores range from 1-4 with highest scores indicating higher self-efficacy. The total score is calculated by finding the sum of the all items.
Feasibility - intervention implementation | up to 6 months post intervention commencement
  Feasibility of Implementation Measure (completed by service leads and clinicians)
Vocational specialist confidence and competence | Immediately post-training
  Purpose-built scale (no title or acronym) developed specifically for the current study capturing self-report vocational specialist confidence and competence using VR for vocational support. The scale is 8 items, scored of a scale of 1 to 4. Higher score indicates a greater degree of competence with VR4VR.
Implementation - perceived barriers and enablers to use in practice | Through study completion an average of 6 months
  Assessed through qualitative analysis of supervision meeting minutes with vocational specialists
Implementation - perceived barriers and enablers to use in practice | Through study completion an average of 6 months
  Assessed through qualitative analysis of research meeting minutes
Implementation - perceived barriers and enablers to use in practice | Through study completion an average of 6 months
  Assessed through qualitative analysis of post-intervention interviews focusing on participants' experiences of using the VR4VR intervention during vocational support.
Feasibility - fidelity | 6 months post intervention commencement
  Proportion of VR4VR sessions that are delivered per-protocol, assessed by the timing of sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Nicholas, PhD, Principal Investigator — University of Melbourne
Locations (3):
- Australia (3):
  - Veritas House, Orange, New South Wales
  - Orygen Specialist Services, Melbourne, Victoria
  - Youth Focus Burswood, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No
Unable to share individual participant data due to restrictions from ethics approval and small exploratory nature of the current trial.